CLINICAL TRIAL: NCT03800888
Title: Real-time Tuberculosis Medication Adherence Intervention in Rural Southwestern Uganda
Acronym: MAT K43
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: Massachusetts General Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUST-16/10-16
Record Dates: First submitted 2019-01-04; First posted 2019-01-11 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Tuberculosis
Keywords: Real-time; Medication Adherence; Tuberculosis
MeSH Terms: conditions — Tuberculosis; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using the 1:1:1 allocation ratio to the following arms: 1) Fixed and linked SMS reminders, 2) SMS notifications to social supporters, and 3) no SMS (control). All participants will have adherence monitored in real-time for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants in Arm A will receive a Wisepill device for Real- time monitoring plus Daily SMS reminders plus Social Supporter notifications (for 3 months) sent according to participant's preferred time and then shall receive Linked SMS for missed dose (Right after missed dose) plus Social Support notifications (3 months).
  Interventions: Other: Daily SMS reminders for TB patients; Other: SMS Notifications for social supporters
- Arm B (Experimental): Participants in Arm B will receive a wisepill device for Real-time monitoring plus Weekly SMS reminders plus Social support notifications (for 3 months) sent according to participant's preferred time and date and then shall receive Linked SMS for missed dose (Right after missed dose) plus Social Support notifications (3 months).
  Interventions: Other: SMS Notifications for social supporters; Other: Weekly SMS remiders
- Arm C (No Intervention): Participants in Arm C will receive only the Wise pill device (No SMS)

INTERVENTIONS:
Other: Daily SMS reminders for TB patients — Daily SMS Medication reminders will be sent to TB patients to remind them take their medications.
  Arms: Arm A
Other: SMS Notifications for social supporters — SMS Notifications will be sent to social supporters to assit TB patients take their medication
  Arms: Arm A; Arm B
Other: Weekly SMS remiders — Weekly SMS reminders sent to TB patients to remind them take medication
  Arms: Arm B

SUMMARY:
With an estimated 60,000 people diagnosed with TB (Tuberculosis) annually, Uganda holds the 16th position of the 22 countries with highest cases of TB in the world. The Uganda national target of utilizing the DOTS (Direct Observed Treatment Short Course) to successfully treat 85% of patients diagnosed with TB has not been met. Currently, the country only detects 49.6% TB case detection, of which it successfully treats 73%. The DOTS strategy has suffered many socioeconomic challenges, which have resulted into its abandonment by many of the Ugandan hospitals. Poor TB medication adherence greatly attribute to the many cases of TB in Uganda. Causes of non-adherence to TB medication include lack of patient follow-up, patients' lack of transport to go to the clinics to pick up drugs, patients' forgetfulness. There is evidence that real time adherence monitoring linked with SMS reminders and social support notifications can address barriers to sustained ART (antiretroviral therapy) adherence. Such novel interventions addressing TB medication adherence challenges in low resource settings to date are limited. The prevailing SMS-based studies for TB medication adherence report mixed results, do not strategically link interventions with missed doses, and have largely been implemented in developed countries. To date, little is known about the use of real-time adherence monitoring technologies for TB medication adherence in resource-limited settings.

The goal of this research is to investigate the use of real time adherence monitoring technology linked with SMS reminders and notifications for TB medication adherence in rural southwestern Uganda.

The investigator will develop and quantitatively test a real-time adherence monitoring intervention with 60 individuals initiating TB treatment, and 40 social supporters. The investigator will randomize participants (1:1:1) to the following arms: 1) Fixed and linked SMS reminders, 2) SMS notifications to social supporters, and 3) no SMS (control). All participants will have adherence monitored in real-time for 6 months.

DETAILED DESCRIPTION:
This study has three major aims (Aims 1, 2 and 3)

Aim 1: Carry out a formative qualitative study to assess barriers and facilitators to TB medication adherence, and identify optimal SMS reminders, notifications, and initial feasibility of real time adherence monitoring. 35 TB patients will be recruited from the TB clinic in Mbarara Regional Referral Hospital (MRRH), and up to 15 social supporters specified by the TB patients (one per TB patient). Drawing from technology adoption and behavioral change models, the investigator will use semi-structured interviews to assess the initial feasibility and acceptability of the intervention, as well the barriers and facilitators to TB medication adherence, and how they can be addressed using the proposed intervention. The purpose will be to inform the development the technology necessary to conduct a real-time intervention involving a wireless monitor and SMS reminders and notifications (Aim 2 and 3).

Aim 2: Develop a TB medication adherence intervention based on SMS reminders (fixed and/or linked to real-time detection of missed doses) and assess its acceptability, feasibility and preliminary impact on adherence.

The Investigators will use real-time electronic adherence monitoring (i.e., Wisepill) to follow 60 TB-infected individuals initiating TB treatment in Mbarara Regional Referral Hospital (MRRH) for six months. Using a 1:1:1 manner, participants will be randomized to one of the following three study arms (details of each intervention will be informed by the data collected in Aim 1):

1. Intervention Arm A: SMS reminders on a fixed schedule
2. Intervention Arm B: SMS reminders linked to missed doses
3. Control: No SMS reminders.

Qualitative interviews to understand the patients experiences with Wisepill adherence monitoring and the SMS reminders will be carried out, depending on the study arm to which they are assigned. The first set of interviews for Arms A and B will be conducted at the end of Month 3 of the study. The second set of interviews is planned to be conducted within two weeks after the first 24+ hour lapse in Wisepill signal for the participants in the intervention arms (A and B). If there is no 24+ hour lapse, the interview will take place at the end of the study. The control participants in Arm C's interview will occur at a convenient time during Months 3-6. The effect sizes will be estimated by comparing adherence at the end of six months between each intervention group and the control group. The primary outcome will be percent adherence.

Treatment outcomes will be defined according to WHO definitions, where cure and completed treatment are defined as successful treatment outcomes (WHO 2014). Unsuccessful treatment outcomes for active TB treatment will include death ascertained from hospital death registry, treatment failure (sputum smear positive at 6 months) and loss to follow-up. Treatment outcomes will be compared for both intervention and control arms.

Aim 3: Develop a social support intervention linked to real-time adherence monitoring and assess its acceptability, feasibility and preliminary impact on adherence. Members of pre-existing social support networks for the same 40 TB-infected individuals in the two intervention arms described in Aim 2 above will be recruited to receive real-time SMS notification of sustained non-adherence (i.e., gaps of >24 hours) over the latter four months of follow-up. The investigators will continue to follow the 20 TB-infected individuals in the control group (i.e., electronic monitoring alone) to estimate the effect size of the intervention on adherence at the end of the six-month period. Qualitative interviews to understand the experiences of participants in each study arm and the social supporters with special emphasis on understanding mechanisms of effects of the SMS reminders, forms and dynamics of support, experiences with the SMS reminders/notifications, and technical problems encountered will be conducted. The results of Aim 3 will be used to determine the types of SMS (fixed versus linked SMS), and the nature of social support that shows the most promise for real time intervention on anti-TB medication adherence and cure.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Wisepill participants:

* Newly diagnosed with TB per the clinic records
* Starting TB treatment now or within the next two weeks
* Age 18 years and older
* Live in the Mbarara District (20 km from MRRH)
* Own a cell phone for personal use and have reliable cellular phone reception at home on networks (MTN or Airtel) supported by the technology used in this study
* Know how to use SMS
* Willing and able to give consent
* Willing and able to name one or two social supporters who are able to use SMS and have cellular phones using network provider (MTN or Airtel) supported by the technology used in this study.

Exclusion Criteria for Wisepill Participants:

* Unable to use SMS (The investigators will train and test this skill at recruitment)
* Unwilling to receive SMS reminder
* Severe mental condition limiting the ability to provide consent
* Cellular phone reception is not reliable

Inclusion Criteria for Social Supporters

* Know a Wisepill participant and be aware s/he has TB
* Have provided help to that Wisepill participant at least once, i.e,

  * Helping him/her get to clinic by loaning or giving money, driving the patient , or taking care of his/her job or children while he/she is away
  * Helping the patient take medicines through encouragement or reminders
  * Motivating the patient to take medicines, including addressing cognitive and behavioral barriers such as depression and alcohol use
* Age 18 years or older
* Live in Mbarara District (within 20 KM from MRRH)
* Willing and able to provide consent.

Exclusion:

* Unable to use SMS (Investigators will train and test this skill at recruitment)
* Unwilling to receive SMS reminder
* Severe mental condition limiting the ability to provide consent
* Cellular phone reception is not reliable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Percent adherence | 12 Weeks
  SPSS (statistical package for social scientists) will be used, to determine the mean (standard deviation), median (interquartile range), number of late doses, number of missed doses, and number of hour gaps in adherence as determined by Wisepill for each stage of the intervention, as well as for the control group. The Investigator will compare adherence during each type of SMS reminder with adherence during the matched time period for the control group using T-tests (or Mann-Whitney U tests, depending on the normality of the data) for continuous data and chi-squared tests for categorical data.

SECONDARY OUTCOMES:
Treatment success rate. | 24 Weeks
  The Investigator will determine the mechanisms of effect and context of an integrated adherence monitoring, SMS reminders and social support interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Musiimenta A. Social and Institutional issues in the Adoption of School-based Technology-aided Sexual Health Education Program. Online J Public Health Inform. 2013 Jul 1;5(2):213. doi: 10.5210/ojphi.v5i2.4654. Print 2013. PMID 23923098
- [Background] Musiimenta A. A Controlled Pre-Post Evaluation of a Computer-based HIV/AIDS Education on Students' Sexual Behaviors, Knowledge and Attitudes. Online J Public Health Inform. 2012;4(1):ojphi.v4i1.4017. doi: 10.5210/ojphi.v4i1.4017. Epub 2012 May 17. PMID 23569630
- [Background] Musiimenta A. Contextual Mediators influencing the Effectiveness of Behavioural Change Interventions: A Case of HIV/AIDS Prevention Behaviours. Online J Public Health Inform. 2012;4(2):ojphi.v4i2.3988. doi: 10.5210/ojphi.v4i2.3988. Epub 2012 Sep 14. PMID 23569636
- [Background] Liu X, Lewis JJ, Zhang H, Lu W, Zhang S, Zheng G, Bai L, Li J, Li X, Chen H, Liu M, Chen R, Chi J, Lu J, Huan S, Cheng S, Wang L, Jiang S, Chin DP, Fielding KL. Effectiveness of Electronic Reminders to Improve Medication Adherence in Tuberculosis Patients: A Cluster-Randomised Trial. PLoS Med. 2015 Sep 15;12(9):e1001876. doi: 10.1371/journal.pmed.1001876. eCollection 2015 Sep. PMID 26372470
- [Background] Nglazi MD, Bekker LG, Wood R, Hussey GD, Wiysonge CS. Mobile phone text messaging for promoting adherence to anti-tuberculosis treatment: a systematic review. BMC Infect Dis. 2013 Dec 2;13:566. doi: 10.1186/1471-2334-13-566. PMID 24295439
- [Derived] Musiimenta A, Tumuhimbise W, Atukunda EC, Mugaba AT, Musinguzi N, Muzoora C, Bangsberg D, Davis JL, Haberer JE. The feasibility, acceptability, and preliminary impact of real-time monitors and SMS on tuberculosis medication adherence in southwestern Uganda: Findings from a mixed methods pilot randomized controlled trial. PLOS Glob Public Health. 2023 Dec 5;3(12):e0001813. doi: 10.1371/journal.pgph.0001813. eCollection 2023. PMID 38051699